CLINICAL TRIAL: NCT01555203
Title: A Multiple Health Behavior Change Internet Program for College Students
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R44HL074485-04 (NIH)
Record Dates: First submitted 2011-08-15; First posted 2012-03-15 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Sedentary Lifestyle; Stress, Psychological; Healthy Eating
MeSH Terms: conditions — Sedentary Behavior; Stress, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- liveWell: A healthy foundation for life (Experimental)
  Interventions: Behavioral: liveWell: A healthy foundation for life

INTERVENTIONS:
Behavioral: liveWell: A healthy foundation for life — liveWell is a unique online, mobile-compatible, multi-media, evidence-based program designed to help college students exercise, eat healthy, and manage stress. At the core of the Transtheoretical Model-based intervention is a computer-tailored behavior change intervention (CTI) that analyzes students' responses to reliable and valid assessments of key behavior change constructs using empirically derived pre-programmed decision rules. The rules determine which feedback users receive on how they are doing compared to their peers in their same stage. At follow-up, feedback is further tailored to how students are doing compared to their last session.
  In addition to the CTI, completed three times during the semester, liveWell includes a dynamic portal that is populated with a variety of engaging and interactive stage-matched activities and resources. The portal provides more content and specifics on how to apply each of the processes and principles of change introduced in the CTI.

SUMMARY:
The objective of this Phase II research is to evaluate the effectiveness of a population-based, individually tailored multiple health behavior change program for exercise, healthy eating, and stress management in a randomized trial including approximately 1,500 college students.

DETAILED DESCRIPTION:
Despite the importance of shaping a solid foundation of health behaviors early in life, college students have been understudied as a population for health promotion programs. This study represents innovative research for impacting the promotion of healthy lifestyles among college students. The objective is to develop and test a population-based, multiple health behavior change program for college students, liveWell: A Healthy Foundation for Life.

The multiple behavior multimedia program will offer Transtheoretical Model-based (TTM) computer tailored feedback on regular exercise, fruit and vegetable consumption, and effective stress management, as well as providing access to a stage-matched dynamic web portal. The TTM is a comprehensive model that integrates ideas from several different theories and approaches to change (hence the name "Transtheoretical") to explain and predict how and when individuals end high-risk behaviors or adopt healthy ones. Thirty years of research has consistently demonstrated that change is a process that unfolds over time through a series of stages: Precontemplation, Contemplation, Preparation, Action, and Maintenance. It matches specific principles and processes of change to each person's stage of change and guides individuals through the change process. The TTM has been applied throughout the world to behaviors such as smoking cessation, alcohol reduction, bullying prevention, weight management, and medication adherence.

A primary goal of this Phase II grant is to assess the effectiveness of liveWell in a randomized trial including 1680 students from 2 large universities in the U.S. Students will be recruited via freshman orientation classes and will complete follow-up assessments at 6-and 12-months. Effectiveness will be assessed by comparing improvements in continuous outcome measures and movement to public health criteria for each behavior. This intervention offers a cost-effective, science-based, and easily deliverable solution to improve multiple health behaviors, and overall health and well-being, of college students.

ELIGIBILITY:
Inclusion Criteria:

* enrolled as a freshmen in college
* English speaking

Exclusion Criteria:

-

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1877 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Adoption of Healthy Eating at 6 & 12 months | Baseline, six months and twelve months
  Continuous measure of fruit and vegetable intake: stage of readiness for fruit and vegetable intake.
Change from Baseline in Adoption of Exercise at 6 & 12 months | Baseline, six months and twelve months
  Godin Leisure Time Exercise Questionnaire and stage of readiness for regular exercise
  Triaxial accelerometers in sub-sample of participants
Change from Baseline in Adoption of Exercise, Healthy Eating, and Effective Change from Baseline in Adoption of Effective Stress Management at 6 & 12 months | Baseline, six months and twelve months
  RISCI: Rhode Island Stress and Coping Inventory and stage of readiness for effective stress management

CONTACTS AND LOCATIONS:
Overall Officials: Sara Johnson, PhD, Principal Investigator — Pro-Change Behavior Systems, Inc.